CLINICAL TRIAL: NCT03712072
Title: Multi-modal Neuroimaging in Children With Cerebral Palsy or Brachial Plexus Birth Palsy to Assess Functional and Anatomical Reorganization in Relation to Sensory and Motor Functions
Brief Title: Multi-modal Neuroimaging in Children With Cerebral Palsy or Brachial Plexus Birth Palsy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Christos Papadelis, Principal Investigator, Boston Children's Hospital
Other Study IDs: IRB-P00023570
Record Dates: First submitted 2018-01-24; First posted 2018-10-19 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Palsy; Brachial Plexus; Injury, Newborn
MeSH Terms: conditions — Cerebral Palsy; Wounds and Injuries | interventions — Magnetoencephalography; Electroencephalography; Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Children with Cerebral Palsy: Data from the participants with Cerebral Palsy will be collected over the course of four visits: (i) the recording session for the Magnetoencephalography (MEG), (ii) the recording session for the Electroencephalography (EEG), (iii) the Magnetic Resonance Imaging (MRI) scanning session, and (iv) the Transcranial Magnetic Stimulation (TMS) session.
  Interventions: Device: Magnetoencephalography (MEG); Device: Electroencephalography (EEG); Device: Transcranial Magnetic Stimulation (TMS)
- Children with BPBP: Data from the participants with Brachial Plexus Birth Palsy will be collected over the course of four visits: (i) the recording session for the Magnetoencephalography (MEG), (ii) the recording session for the Electroencephalography (EEG), (iii) the Magnetic Resonance Imaging (MRI) scanning session, and (iv) the TMS session.
  Interventions: Device: Magnetoencephalography (MEG); Device: Electroencephalography (EEG); Device: Transcranial Magnetic Stimulation (TMS)
- Typically Developing Children: Data from the typically developing participants will be collected over the course of four visits: (i) the recording session for the Magnetoencephalography (MEG), (ii) the recording session for the Electroencephalography (EEG), (iii) the Magnetic Resonance Imaging (MRI) scanning session, and (iv) the Transcranial Magnetic Stimulation (TMS) session.
  Interventions: Device: Magnetoencephalography (MEG); Device: Electroencephalography (EEG); Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Magnetoencephalography (MEG) — The purpose of the device is to measure magnetic fields produced by an individual's brain and provide information on the location of the source of the fields. Participants between the ages of 0-3 years of old whose head can fit in the MEG helmet will be the patient population used for the BabyMEG. The device will be used in this study to learn more about the somatosensory and motor networks of children who have cerebral palsy and compare their brain signals to healthy children.
  Other Names: MagView Biomagnetometer
Device: Electroencephalography (EEG) — The device is an EEG cap - a non-invasive EEG positioning system used to quickly place a large number of surface electrodes in a quick and consistent manner on the head. The device will measure electrophysiological signals from the scalp.
  Other Names: Waveguard (TM) EEG cap
Device: Transcranial Magnetic Stimulation (TMS) — The device will be used for motor mapping. Motor threshold is operationally defined as minimum machine output necessary to elicit a response from the abductor pollicis brevis right (APB), contralateral to the stimulated hemisphere, of 50 microvolts, on >50% of trials. Upper limb motor mapping is conducted at 110% abductor pollicis brevis motor threshold in each hemisphere, or at 100% machine output (MO). Lower limb motor mapping is conducted at a fixed machine output corresponding to the magnitude sufficient to elicit reliable tibialis anterior (TA) motor evoked potentials (MEPs). Single pulse TMS is performed while motor evoked potentials are recorded bilaterally from the APB, deltoid, and TA using surface electromyography (EMG).
  Other Names: Nexstim Navigated Brain Stimulation (NBS) System 4

SUMMARY:
The main goal of this study is to identify abnormal functional and anatomical brain reorganization associated with hand, foot, and shoulder function in children (0-18 years old) with cerebral palsy (CP) due to periventricular white matter injury (PV-WMI) or brachial plexus birth palsy (BPBP) using a multi-modal neuroimaging approach.

DETAILED DESCRIPTION:
This is a non-interventional study designed to assess changes in the sensorimotor cortex of children with CP as a result of PV-WMI and children with BPBP that combines multiple neuroimaging techniques to better visualize the resulting brain reorganization. The study design will be a mixed 3 (group: CP, BPBP, TD) x 2 (hemisphere: more affected, less affected) analysis of variance (ANOVA), with group being a between-subject factor and hemisphere a within-subjects factor.

The research study plans to recruit and test 30 children with CP due to PV-WMI, 30 children with BPBP, and 30 aged-matched and typically developing (TD) children aged from 0 to 18 years old.

Data from the participants will be collected over the course of four visits: (i) the recording session for the MEG, (ii) the recording session for the EEG, (iii) the MRI scanning session, and (iv) the TMS session. TD, CP, and BPBP subjects will be asked to commit to these visits.

The MEG session will last ~3 hours with the actual measurements lasting ~60 minutes, the EEG session will last ~2 hours with the actual measurements lasting ~60 minutes, the MRI visit will last ~1 hour with the actual acquisition scan timing lasting ~30 minutes, and the TMS visit will last ~1 and a half hours with the actual acquisition time lasting ~45 minutes. Depending on the participant, the behavioral tests may be administered during any of the visits that the child is most comfortable and able to perform them.

ELIGIBILITY:
Inclusion Criteria:

Children with Cerebral Palsy should have:

* An evaluation by a pediatric neurologist with a diagnosis of CP due to PV-WMI,
* Absence of any genetic syndrome diagnosis,
* No history of trauma or brain operation,
* Classified as high-functioning (I or II) at the Gross Motor Function Classification System (GMFCS)32.

Children with Brachial Plexus Birth Palsy should have:

* An evaluation by a hand and upper extremity surgeon with a diagnosis of BPBP
* May or may not have undergone primary microsurgical or secondary reconstructive operations prior to this study.

Typically Developing children should have:

* No history of neurological disorder or brain injury.

Exclusion Criteria:

Children will be excluded if they meet any of the follow criteria, determined via their medical and developmental history:

* Having a hard time sitting still,
* Presence of any metal implants,
* Baclofen pumps,
* History of traumatic brain injury or brain operation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children (0-18 years old) with cerebral palsy (CP) due to periventricular white matter injury (PV-WMI) or brachial plexus birth palsy (BPBP) using a multi-modal neuroimaging approach.
  The investigators plan to recruit and test 30 children with CP due to PV-WMI, 30 children with BPBP, and 30 aged-matched and typically developing (TD) children aged from 0 to 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Somatosensory evoked potentials as assessed using MEG | Approximately two years
  The amplitude of somatosensory evoked fields (in fempto-Tesla) at the peak of the first cortical response after tactile stimulation will be measured and reported for each stimulation site, each hemisphere & each patient.

SECONDARY OUTCOMES:
Motor evoked amplitude as assessed using MEG | Approximately two years
  The amplitude of motor evoked fields (in fempto-Tesla) at the peak of the first cortical response after finger movement will be measured and reported for each site, each hemisphere & each patient.
Somatosensory evoked potentials as assessed using EEG | Approximately two years
  The amplitude of somatosensory evoked potentials (in micro-Volts) at the peak of the first cortical response after tactile stimulation will be measured and reported for each stimulation site, each hemisphere & each patient.
Motor evoked potentials as assessed using EEG | Approximately two years
  The amplitude of motor evoked potentials (in micro-Volts) at the peak of the first cortical response after finger movement will be measured and reported for each site, each hemisphere & each patient.
Cortical excitability of motor cortex assessed using TMS | Approximately two years
  The resting motor threshold (Volts/meter) of the primary motor cortex will be measured and reported for each hemisphere & each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Papadelis, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States